CLINICAL TRIAL: NCT04649645
Title: International Randomized Controlled Trial Evaluating Changes in Oral Health in Smokers After Switching to Combustion-Free Nicotine Delivery Systems: SMILE Study Protocol
Brief Title: Changes in Oral Health in Tobacco Cigarettes Smokers After Switching to Combustion-Free Nicotine Delivery Systems
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eclat Srl. (Other)
Collaborators: University of Catania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: COE1-05-SMILE
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Gingivitis; Periodontal Diseases
Keywords: Electronic cigarettes; Tobacco Harm Reduction; Heated tobacco products; Smokers; Gingivitis; Modified gingival index; Oral Health; Tooth stain; Periodontitis; Dental plaque imaging; Dental discoloration
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Vaping; Tooth Discoloration; Periodontitis | interventions — Tobacco Products

STUDY DESIGN:
Intervention Model Description: Smokers participants who were eligible and consent to take part will be randomized to either continuing smoking their own cigarette brand (Arm A) or switching to using C-F NDS (Arm B). Never-smokers participants who were eligible and consent to take part will be assigned to Arm C.
  The randomization sequence will be computer generated, with an allocation ratio of 1:4 (Study Arm A : Study Arm B; Smokers : N-C NDS users) to compensate for an estimated 25% success rate (combined smoking abstinence rate + >90% smoking reduction rate) in the long term. The randomization scheme will be provided to clinical sites via a web-based application set up by the CRO. The staff randomizing the participant will access the web-based application when the participant is with them, entering their participant identification number, date of birth and initials into the program. The allocation will be immediately provided by the program/software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard Arm (Arm A) (Active Comparator): Participant continues smoking their own cigarette brand.
  Interventions: Other: TOBACCO CIGARETTES
- Intervention Arm (Arm B) (Active Comparator): Participant switches to using C-F NDS.
  Interventions: Other: COMBUSTION-FREE NICOTINE DELIVERY SYSTEMS (C-F NDS)
- Control Arm (Arm C) (Active Comparator): Participant continues to not smoking or using of any nicotine/tobacco products.
  Interventions: Other: NOT SMOKING

INTERVENTIONS:
Other: TOBACCO CIGARETTES — Participants in Arm A will continue smoking their own cigarette brand as usual.
  Arms: Standard Arm (Arm A)
Other: COMBUSTION-FREE NICOTINE DELIVERY SYSTEMS (C-F NDS) — Participants in Arm B will trial and familiarize with a selection of C-F NDS in order to choose the product of their preference. They will be trained and counselled on the chosen C-F NDS. Prior to check-out, participants wishing to use a heated tobacco device will receive one kit and a full 2 weeks supply of tobacco sticks of their choice (they will receive a number of tobacco sticks per day corresponding to the number of cigarettes smoked at baseline); those wishing to use a vaping product will receive one vaping kit and a full 2 weeks supply of e-liquids of their choice (they will receive twelve 10 ml refill containers).
  Arms: Intervention Arm (Arm B)
Other: NOT SMOKING — Participants in Arm C will continue not smoking or use any form of tobacco or nicotine-containing products.
  Arms: Control Arm (Arm C)

SUMMARY:
Although the well-known detrimental effects of conventional cigarette smoking on oral health, there are still lack of evidences about the impact of less harmful alternatives (such as electronic cigarettes or heat not burn products), especially in young smokers with clinical absence of signs of moderate to severe periodontitis.

This study aims to investigate whether cigarette smokers who switch to combustion-free nicotine delivery systems (C-F NDS) undergo measurable improvements in oral health parameters and teeth appearance, comparing short- and long-term impact on periodontal health between smokers continuing with conventional cigarette smoking, those switching to combustion-free nicotine delivery systems (C-F NDS), and never-smokers.

The investigator propose a prospective, multicenter, interventional, open label, randomized, controlled, three parallel-arms study assessing oral health parameters and teeth appearance of 18 months duration.

DETAILED DESCRIPTION:
SMILE is an international, open label, randomized, controlled study of 18 months duration designed to assess whether cigarette smokers switching to combustion free-nicotine delivery systems (C-F NDS) will undergo measurable improvements in oral health parameters and teeth appearance as a consequence of avoiding exposure to cigarette smoke. Five countries have so far agreed to participate: Italy, Moldova, Poland, UK and Indonesia. An amendment will be submitted to the REC once the final two countries are signed up.

A volunteer population of never-smokers and regular smokers of conventional cigarettes with a clinical absence of signs of periodontitis will be recruited. Regular cigarette smokers will be randomized 1:4 ratio either continuing to smoke commercially manufactured conventional cigarettes (Study Arm A) or switching to C-F NDS (Study Arm B). Never Smokers will be assigned to Arm C.The intended minimum number of participants by the end of the study is 460.

Before randomization, all smokers will be reminded of the risks associated with smoking and will be offered a free smoking cessation program according to standard local guidelines and depending on the local availability of antismoking services. Those who decline the invitation will be eligible for recruitment into the study.

Smokers are free to voluntarily quit smoking/C-F NDS and/or withdraw from the study at any time.

Duration:

All participants will attend a total of seven clinics visits: Day -28 to Day -1 - Screening; Day 0 - Enrollment and Randomization (Visit 0); Day 14 (+/-3 days) - Baseline Visit (Visit 1); Day 90 (+/-5 days) - Visit 2; Day 180 (+/-7 days) - Visit 3; Day 360 (+/-10 days) - Visit 4; Day 540 (+/-10 days) - Visit 5.

Each participant will undergo screening within 28 days prior to Visit 0. Eligible participants will be enrolled and randomized on Visit 0. Baseline assessments will be performed at Visit 1, 14 days after Visit 0. The overall duration of study participation for each participant will be a maximum of 568 +/- 10 days.

The randomization sequence will be computer generated, with an allocation ratio of 1:4 (Study Arm A : Study Arm B; Smokers : N-C NDS users) to compensate for an estimated 25% success rate (combined smoking abstinence rate + >90% smoking reduction rate) in the long term. The randomization scheme will be provided to clinical sites via a web-based application set up by the CRO. The staff randomizing the participant will access the web-based application when the participant is with them, entering their participant identification number, date of birth and initials into the program. The allocation will be immediately provided by the program/software.

Product use Regular smokers will continue to smoke their usual brand of conventional cigarette until Baseline on Visit 1. After Visit 1, participants on both Arms A and B will be asked to use only their assigned products ad libitum for the whole duration of the study.

Participants in Arm A will continue smoking their own conventional cigarette brand, as usual.

Participants in Arm B will have the option to try and choose among a selection of either three e-liquids or three tobacco sticks (depending on the C-F NDS they have chosen). They will also be trained and instructed on how to correctly use their chosen C-F NDS. Participants wishing to use a heated tobacco device (HTD) will receive the number of tobacco sticks per day corresponding to the number of cigarettes smoked per day at baseline. Participants wishing to use a vaping product will receive one vaping kit and supply of e-liquids of their choice enough to provide consumption in between supply visits (see Table 2); on average they will receive 4 x 10 ml refill containers per week. Free products will be supplied at each subsequent visit throughout the whole duration of the study.

Participants in Arm C will continue to not smoking or use any form of tobacco or nicotine-containing products.

A prospective monitoring of cigarette consumption, C-F NDS use, and oral hygiene routine will be carried out throughout the study with the tracker APP. Moreover, participants in Arm B will be asked to return all empty, part-used, and unused consumables (tobacco sticks, e-cigarette cartridges, e-liquid refill bottles) at each study visit.

Justification for Study Design

Participants in this study will be a minimum of 18 years of age. This is based on:

* The legal age to obtain tobacco products is 18 years
* The presence of at least 10 natural anterior permanent teeth in total (cuspid to cuspid, lower and upper jaw).

To investigate the effects of abstaining from smoking by switching in smokers with clinical absence of periodontitis, a population of both smokers who are intending to make the switch to N-C NDS and never-smokers will be recruited. By the end of the study, it is estimated that a high proportion (approx. 75%) of patients randomized in the Arm B of the study will not be able to achieve success (defined as either complete smoking abstinence or as at least 90% smoking reduction). To account for this, the C-F NDS population will be over sampled and a 1:4 randomization ratio scheme (i.e. for every patient randomized in the continue-to-smoke population, four will be randomized in the C-F NDS population) will be adopted.

It will not be possible to blind participants to the intervention they will be receiving. It will not be possible to blind trial staff when providing the interventions and collecting data. However, data analyses will be conducted blind to Study Arms allocation. All other trial staff who have access to outcome data will remain blinded until prespecified data analyses will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrate understanding of the study and willingness to participate in the study by providing a signed written informed consent
* Healthy subjects, not taking regular medications for chronic medical conditions
* Adults, age at least 18 years old.
* Presence of at least 10 natural anterior teeth in total (cuspid to cuspid, lower and upper jaw).
* Presence of at least 18 'scorable' teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, orthodontically banded, exhibiting general cervical abrasion and/or enamel abrasion, and third molars will not be included in the tooth count;
* Willingness and ability to comply with the requirements of the study including installing an APP on their digital device, e.g. smart phone or tablet.

For Arms A and B, subject have to be:

* Regular smokers, defined as:

  * Smoked for at least five consecutive years prior to Screening.
  * Smoked >10 and < 30 cigarettes per day (CPD).
  * with an exhaled breath carbon monoxide (CO) level ≥7 ppm at Screening.
* willing to regularly use of any nicotine or tobacco product other than their own conventional cigarettes brand within 14 days prior to Screening.
* willing to change to use of study products or if randomized to Arm A continuing to use their own brand of conventional cigarettes for the whole duration of the study.

For Arm C, subjects have to be:

* Never-smokers, defined as:

  * never smoked or who have smoked < 100 cigarettes in their lifetime and none in the 30 days prior to screening.
  * with an exhaled breath CO level < 7 ppm at screening.
* willing to not smoke or use any form of tobacco or nicotine-containing products for the whole duration of the study.

Exclusion Criteria:

* Pregnancy.
* Presence of extensive crown or bridge work, dental implants, and/or rampant decay (per Investigator/Examiner discretion)
* Significant oral soft tissue pathology or any type of gingival overgrowth, other than plaque-induced gingivitis and mild periodontitis (Stage I)
* Moderate to Severe Periodontitis (Stage II, III and IV) based on 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions, which require:

  * Detectable Interdental Clinical Attachment Loss (CAL) ≥ 3 mm at ≥ 2 non-adjacent teeth.
  * Buccal or Oral CAL ≥3 mm with pocketing ≥ 5 mm detectable at ≥ 2 teeth.
* Removable dentures or fixed and removable orthodontic appliance (except fixed lingual wires).
* Significant history of alcoholism or drug abuse (other than tobacco/nicotine) within 24 months prior to screening, as determined by the Investigator.
* A course of treatment with any medications or substances (other than tobacco/nicotine) which:

  * interfere with the cyclooxygenase pathway (e.g. anti-inflammatory drugs including aspirin and ibuprofen) within 3 days prior to each visit.
  * are known to have antibacterial activity (e.g. antibiotics) within 7 days prior to each visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Modified Gingival Index (MGI) | Changes in the severity of gingivitis from baseline will be assessed at 3 months, 6 months, 12 months and 18 months
  Percentage (%) mean changes in MGI from baseline at different study time-points

SECONDARY OUTCOMES:
Macpherson Modification of Lobene Tooth Stain Index (MLSI) | Changes in extent and severity of tooth stains from baseline will be assessed at 3 months, 6 months, 12 months and 18 months
  Change in MLSI from baseline at different study time-points
Dental Discolorations | Changes in dental discolouration from baseline will be assessed at 3 months, 6 months, 12 months and 18 months
  Percentage (%) mean change in dental shade (L, a*, b*) from baseline at different study time-points
Plaque Score Imaging (QLF) | Changes in dental plaque from baseline will be assessed at 3 months, 6 months, 12 months and 18 months
  Changes in ΔR30 and ΔR120 from baseline at different study time-points
Oral Health Quality of Life (OHQOL) | Changes in OHQOL score from baseline will be assessed at 3 months, 6 months, 12 months and 18 months
  Changes in OHQOL from baseline at different study time-points
EuroQoL Visual Analog Scale (EQ VAS - QoL) | Changes in the EQ VAS - QoL score from baseline will be assessed at 3 months, 6 months, 12 months and 18 months
  Changes in EQ VAS-QoL from baseline at different study time-points

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pacino, D.D.S., Principal Investigator — Addendo srl, Catania, Italy
Locations (1):
- Addendo srl, Catania, Catania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Offenbacher S. Periodontal diseases: pathogenesis. Ann Periodontol. 1996 Nov;1(1):821-78. doi: 10.1902/annals.1996.1.1.821. No abstract available. PMID 9118282
- [Background] Research, Science and Therapy Committee. Position Paper: Diagnosis of Periodontal Diseases. J Periodontol. 2003 Aug;74(8):1237-1247. doi: 10.1902/jop.2003.74.8.1237. PMID 29539063
- [Background] Armitage GC. Clinical evaluation of periodontal diseases. Periodontol 2000. 1995 Feb;7:39-53. doi: 10.1111/j.1600-0757.1995.tb00035.x. No abstract available. PMID 9567929
- [Background] Czesnikiewicz-Guzik M, D'Aiuto F, Deanfield JE. Understanding residual inflammatory risk sheds new light on the clinical importance of periodontitis in cardiovascular disease. Eur Heart J. 2020 Feb 14;41(7):818-819. doi: 10.1093/eurheartj/ehaa107. No abstract available. PMID 32058578
- [Background] Armitage GC. Periodontal infections and cardiovascular disease--how strong is the association? Oral Dis. 2000 Nov;6(6):335-50. doi: 10.1111/j.1601-0825.2000.tb00126.x. PMID 11355266
- [Background] Bergstrom J. Cigarette smoking as risk factor in chronic periodontal disease. Community Dent Oral Epidemiol. 1989 Oct;17(5):245-7. doi: 10.1111/j.1600-0528.1989.tb00626.x. PMID 2791514
- [Background] Bergstrom J, Preber H. Tobacco Use as a Risk Factor. J Periodontol. 1994 May;65(5):545-550. doi: 10.1902/jop.1994.65.5.545. PMID 29539746
- [Background] Haber J. Smoking is a major risk factor for periodontitis. Curr Opin Periodontol. 1994:12-8. PMID 8032453
- [Background] Bergstrom J. Tobacco smoking and chronic destructive periodontal disease. Odontology. 2004 Sep;92(1):1-8. doi: 10.1007/s10266-004-0043-4. PMID 15490298
- [Background] Ueno M, Ohara S, Sawada N, Inoue M, Tsugane S, Kawaguchi Y. The association of active and secondhand smoking with oral health in adults: Japan public health center-based study. Tob Induc Dis. 2015 Jul 29;13(1):19. doi: 10.1186/s12971-015-0047-6. eCollection 2015. PMID 26225132
- [Background] Eriksen HM, Nordbo H. Extrinsic discoloration of teeth. J Clin Periodontol. 1978 Nov;5(4):229-36. doi: 10.1111/j.1600-051x.1978.tb01916.x. PMID 363748
- [Background] Christen AG. The impact of tobacco use and cessation on oral and dental diseases and conditions. Am J Med. 1992 Jul 15;93(1A):25S-31S. doi: 10.1016/0002-9343(92)90624-k. PMID 1497000
- [Background] Zhu S, Melcer T, Sun J, Rosbrook B, Pierce JP. Smoking cessation with and without assistance: a population-based analysis. Am J Prev Med. 2000 May;18(4):305-11. doi: 10.1016/s0749-3797(00)00124-0. PMID 10788733
- [Background] West R, Zhou X. Is nicotine replacement therapy for smoking cessation effective in the "real world"? Findings from a prospective multinational cohort study. Thorax. 2007 Nov;62(11):998-1002. doi: 10.1136/thx.2007.078758. Epub 2007 Jun 15. PMID 17573444
- [Background] Polosa R, Farsalinos K, Prisco D. Health impact of electronic cigarettes and heated tobacco systems. Intern Emerg Med. 2019 Sep;14(6):817-820. doi: 10.1007/s11739-019-02167-4. Epub 2019 Aug 14. No abstract available. PMID 31414334
- [Background] Polosa R, Rodu B, Caponnetto P, Maglia M, Raciti C. A fresh look at tobacco harm reduction: the case for the electronic cigarette. Harm Reduct J. 2013 Oct 4;10:19. doi: 10.1186/1477-7517-10-19. PMID 24090432
- [Background] Farsalinos KE, Polosa R. Safety evaluation and risk assessment of electronic cigarettes as tobacco cigarette substitutes: a systematic review. Ther Adv Drug Saf. 2014 Apr;5(2):67-86. doi: 10.1177/2042098614524430. PMID 25083263
- [Background] McNeill A, Brose L S, Calder R, Bauld L and Robson D. Evidence review of e-cigarettes and heated tobacco products 2018. A report commissioned by Public Health England.
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Derived] Conte G, Pacino SA, Urso S, Greiling D, Caponnetto P, Pedulla E, Generali L, Consolo U, Checchi V, Gospodaru S, Bordeniuc G, Fala V, Kowalski J, Nowak M, Gorska R, Amaliya A, Chapple I, Milward M, Maclure R, Nardi GM, Polosa R. Changes in Oral Health and Dental Esthetic in Smokers Switching to Combustion-Free Nicotine Alternatives: Protocol for a Multicenter and Prospective Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 23;13:e53222. doi: 10.2196/53222. PMID 38393754
- [Derived] Conte G, Amaliya A, Gupta S, Emma R, Gospodaru S, Bordeniuc G, Fala V, Pacino SA, Urso S, Zucchelli G, Polosa R. Repeatability of dental plaque quantitation by light induced fluorescence technology in current, former, and never smokers. BMC Oral Health. 2023 Jul 13;23(1):480. doi: 10.1186/s12903-023-03154-0. PMID 37443061
- [Derived] Conte G, Pacino SA, Urso S, Emma R, Pedulla E, Cibella F, Stefanini M, Zucchelli G, Polosa R. Repeatability of dental shade by digital spectrophotometry in current, former, and never smokers. Odontology. 2022 Jul;110(3):605-618. doi: 10.1007/s10266-022-00692-x. Epub 2022 Mar 10. PMID 35266059